CLINICAL TRIAL: NCT07334054
Title: Effect of Vitamin D and Branched-chain Amino Acids on Physical Performance and Biomarkers of Muscle Fatigue in Runners: an 8-week Randomized, Double-blind
Brief Title: Effect of Vitamin D and Branched-chain Amino Acids on Physical Performance and Biomarkers of Muscle Fatigue in Runners
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pedro Julian Flores Moreno (Other)
Collaborators: Claudia Ivette Gamboa Gomez (Unknown); Fabian Rojas Larios (Unknown)
Responsible Party: Sponsor-Investigator, Pedro Julian Flores Moreno, Doctor of Medical Sciences, Universidad de Colima
Organization: Universidad de Colima (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2025-15b
Record Dates: First submitted 2025-11-17; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult Male; Runners
MeSH Terms: interventions — Amino Acids, Branched-Chain; Vitamin D; P-2

STUDY DESIGN:
Intervention Model Description: In clinical trial types based on their methodology, this protocol is considered a randomized controlled clinical trial. Based on the behavior of its groups, the research is categorized as a parallel group.
Who Masked: Participant, Investigator
Masking Description: The research is categorized as double-blind parallel groups, the study subjects will be blinded, by not recognizing that they are under supplementation and secondly the principal investigator will also be unaware of the assigned treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (TP + BCAA + VitD) (Experimental): Training Program + Branched-Chain Amino Acids + Vitamin D
  Interventions: Other: Training program; Dietary Supplement: Branched-Chain Amino Acids; Dietary Supplement: Vitamin D
- Group 2 (TP + BCAA + P2) (Experimental): Training Program + Branched-Chain Amino Acids + Placebo 2
  Interventions: Other: Training program; Dietary Supplement: Branched-Chain Amino Acids; Other: Placebo 2
- Group 3 (TP + VitD + P1) (Experimental): Training Program + Vitamin D (1000 IU) + Placebo 1
  Interventions: Other: Training program; Dietary Supplement: Vitamin D; Other: Placebo 1
- Group 4 (TP + P1+ P2) (Placebo Comparator): Training Program + Placebo1 + Placebo 2
  Interventions: Other: Training program; Other: Placebo 1; Other: Placebo 2

INTERVENTIONS:
Other: Training program — Aerobic training program (60-90% of maximum aerobic speed)
  Other Names: TP
Dietary Supplement: Branched-Chain Amino Acids — Branched-chain amino acids (5 gr/day)
  Other Names: BCAA
  Arms: Group 1 (TP + BCAA + VitD); Group 2 (TP + BCAA + P2)
Dietary Supplement: Vitamin D — Vitamin D (1000 IU/day)
  Other Names: VitD
  Arms: Group 1 (TP + BCAA + VitD); Group 3 (TP + VitD + P1)
Other: Placebo 1 — Placebo 1 (5gr/day)
  Other Names: P1
  Arms: Group 3 (TP + VitD + P1); Group 4 (TP + P1+ P2)
Other: Placebo 2 — Placebo 2 (1 tablet/day)
  Other Names: P2
  Arms: Group 2 (TP + BCAA + P2); Group 4 (TP + P1+ P2)

SUMMARY:
Muscle fatigue caused by physical training is understood as a condition related to the inability to maintain action potential, derived from the alteration in skeletal muscle homeostasis. In long-distance recreational runners, prolonged physical work is performed while maintaining the level of intensity, where a level of fatigue intervenes, which overlaps and generates tiredness to execute the movement continuously. In the last 10 years, sports supplementation has been explored as an aid to increase physical performance, improve muscle recovery and prevent sports injuries.

DETAILED DESCRIPTION:
Objective:

To analyze the effects of an 8-week training program (TP) with vitamin D and branched-chain amino acids (BCAA) supplementation on physical performance and biomarkers of muscle fatigue in long-distance recreational runners.

Materials and methods:

An 8-week randomized controlled clinical trial. Participants will be 64 men aged 25 to 44 years, distributed into 4 intervention groups. Group A: Training + BCAA + Vitamin D. Group B: Training + BCAA + Placebo. Group C: Training + Vitamin D + Placebo. Group D: Training + Placebo + Placebo. Biomarkers of muscle fatigue Interleukin 6 (L-6), Creatine Kinase (CK), Lactate (Lact), Testosterone and Cortisol ratio and serum vitamin D (25(OH)D) and physical performance will be assessed by estimating Maximal oxygen consumption (VO2max) and (Maximal aerobic speed) MAS.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25 to 44
* Men
* Agree to participate in the study
* Sign a consent form
* Experience in long-distance running

Exclusion Criteria:

* Have a previous diagnosis of liver disease, asthma, hypertension, diabetes, cancer, anemia
* Have a previous diagnosis of a neurological disorder (Alzheimer's disease, Parkinson's disease, epilepsy)
* Have a musculoskeletal disability
* Be on medication or supplementation
* Hypervitaminosis D (>100 ng/mL)
* Be on a structured training program
* Use anabolic steroids

Ages: 25 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in lactate levels compared to the placebo group | 8 weeks
  mMol/L
Changes in interleukin-6 levels compared to the placebo group | 8 weeks
  pg/ml
Changes in cratine kinase levels compared to the placebo group | 8 weeks
  U/L
Changes in testosterone cortisol ratio compared to the placebo group | 8 weeks
  mcg/dL
Changes in maximal aerobic speed compared to the placebo group | 8 weeks
  km/h
Changes in maximal oxygen consumption compared to the placebo group | 8 weeks
  ml.O2.kg/min

CONTACTS AND LOCATIONS:
Overall Officials: Pedro J Flores Moreno, Doctor of Medical Sciences, Study Director — Universidad de Colima
Locations (1):
- Universidad de Colima, Colima, Colima, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Results and analysis will be shared with other researchers collaborating on the research project.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Ades AE, Kazantzis G. Lung cancer in a non-ferrous smelter: the role of cadmium. Br J Ind Med. 1988 Jul;45(7):435-42. doi: 10.1136/oem.45.7.435. PMID 3395580
- [Background] Tomaszewska H, Lech H, Parcheta B, Piontek E, Wisniewski L. Prader-Willi syndrome in a girl with 47,XX + mar karyotype. Klin Padiatr. 1982 Sep-Oct;194(5):328-31. doi: 10.1055/s-2008-1033832. No abstract available. PMID 7144051